CLINICAL TRIAL: NCT06030076
Title: A Non-interventional, Prospective Cohort, Multicentre, Real-world Evidence Study to Assess the Effects of Switching From a Biologic Treatment to Tildrakizumab Using Patient-reported Outcomes in Adult Participants With Moderate to Severe Plaque Psoriasis in Austria and Switzerland
Brief Title: A Study to Assess the Effects of Switching From a Biologic Treatment to Tildrakizumab Using Patient-reported Outcomes in Adult Participants With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: SW-ATCH
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Tildrakizumab; Moderate-to-severe plaque psoriasis; Prospective
MeSH Terms: conditions — Psoriasis | interventions — tildrakizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tildrakizumab: Participants who have been prescribed tildrakizumab to manage moderate-to-severe plaque psoriasis according to summary of product characteristic (SmPC) in routine clinical practice settings will be observed prospectively for up to 28 weeks.
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — As provided in real-world clinical practice.
  Other Names: Ilumetri®

SUMMARY:
The main aim of this study is to assess the effects of switching from another biologic to tildrakizumab on patient-reported outcomes and to assess psoriasis intensity, patient's quality of life prior and after switching and the individual rationales for switching biologics.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. >=18 years of age.
3. Moderate-to-severe plaque psoriasis currently treated with a biologic therapy (TNFα antagonist, IL12/23 antagonist, IL17 antagonist).
4. Switch to tildrakizumab due to:

   1. primary or secondary treatment failure (PASI >= 3 or ΔPASI < 75 and/or DLQI > 5)
   2. adverse events, contraindication, intolerance
   3. patient wish (dosing regimen), lack of adherence, or other, including nonmedical reason
5. Treatment with tildrakizumab planned in the frame of clinical practice.

Exclusion Criteria:

1. Patient appears to be unwilling or unable to comply with the requirements of the study or who, in the opinion of the Investigator, should not participate in the study.
2. >=3 previous biologic treatments in the last 3 years.
3. Participation in a clinical trial simultaneous to participation in SW-ATCH.
4. Any condition preventing prescription of Tildrakizumab according to the SmPC, including but not restricted to any contraindication or history of hypersensitivity or intolerance.
5. Patient dependent on the Investigator.
6. Previous treatment with Tildrakizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female participants with moderate to severe plaque psoriasis will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire for Medication-11 (TSQM-11) Score | Baseline, Week 28
  TSQM 11-item scale is derived from the TSQM version 1.4, which comprises four domains: global satisfaction, medication effectiveness, convenience, and side effects with scores at each domain ranging from 0 to 100. Higher scores indicating greater satisfaction and lower scores reflecting room for improvement.
World Health Organisation Well-Being Index (WHO-5) Score | Baseline up to Week 28
  The WHO-5 consists of 5-items that measure current mental well-being. Each item is rated on 6-point Likert scale, ranging from 0 (at no the time) to 5 (all of the time). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

SECONDARY OUTCOMES:
Change from Baseline in absolute Psoriasis Area and Severity Index (PASI) Score | Baseline, Week 4, 16 and 28
  The PASI is a measure of psoriasis and psoriatic arthritis severity that will be assessed at baseline and all follow-up visits for participants with psoriasis or psoriatic arthritis. This common clinical measure selects a representative area of psoriasis for each body region. The intensity of redness, thickness, and scaling of the psoriasis is assessed by the clinician. PASI scores range from 0 to 72, with higher scores indicating worse symptoms.
Change from Baseline in Physician's Global Assessment (PGA) Score | Baseline, Week 4, 16 and 28
  The PGA is an instrument used in clinical trials to rate the severity of psoriasis. It is a 5-point scale measurement ranging from 0 to 4, where 0- clear, 1- almost clear, 2- mild, 3- moderate and 4- severe; based on degree of plaque thickening, scaling and erythema.
Change from Baseline in Dermatology Life Quality Index (DLQI) Score | Baseline, Week 4, 16 and 28
  The DLQI consists of 10 items addressing the subject's perception of the impact of their skin disease on different aspects of their quality of life. Each item is scored on a 4-point Likert scale (0 = 'not at all / not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much'). DLQI scores range from 0 to 30, with higher scores indicating worse quality of life.
Number of Participants with Individual Reasons for Initiating Switch to Tildrakizumab | At Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Gesundheitszentrum Citypark Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No